CLINICAL TRIAL: NCT02483065
Title: Impact of Hospital Admission on Patients With Dementia
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hospital Galdakao-Usansolo (Other Government)
Collaborators: Department of Health, Basque Country, Spain (Unknown)
Responsible Party: Principal Investigator, Josune Martin Corral, PhD, Hospital Galdakao-Usansolo
Other Study IDs: 2012111139
Record Dates: First submitted 2015-06-18; First posted 2015-06-26 (Estimated); Last update posted 2015-06-26 (Estimated); Status verified 2015-06

CONDITIONS: Dementia
Keywords: dementia; hospital admission; mortality; health-related quality of life; activities of daily living
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- inpatients with dementia
  Interventions: Other: mortality at discharge and 3-months after the admission in patients with and without dementia
- inpatients without dementia
  Interventions: Other: mortality at discharge and 3-months after the admission in patients with and without dementia

INTERVENTIONS:
Other: mortality at discharge and 3-months after the admission in patients with and without dementia — Patients diagnosed of dementia who ingresed the hospital were informed of the goals of the study and invited to voluntarily participate. In order to take part in the study, patients were required to provide informed consent. All participants were first screened with the Alzheimer's Disease Test. A diagnosis of dementia was generated by an independent clinician experienced in old age psychiatry using a structured clinical assessment based on operationalized DSM-IV criteria. Clinical data were gathered from hospital notes. Information on sociodemographic data, premorbid basic and instrumental activities of daily living, quality of life and burden of the caregiver was gathered from carers and review of hospital notes. In both cohorts, participants were telephoned 3 months after hospital admission to respond the follow-up questionnaires. Patients who decided not to answer them were considered lost to follow-up. All information was kept confidential.

SUMMARY:
People with dementia have complex medical, social, and psychological needs and can be exacerbated by physical illness and the complex relationships between health care systems, patients and their families or caregivers. They are a vulnerable and fragile population that differs significantly from the population without dementia. Therefore, the investigators propose the following objectives: 1. To describe the evolution of dementia patients admitted during the study period in two hospitals in the Basque Health Service-Osakidetza and complications associated with such admissions. 2. To compare with a control group (matched by type of pathology, age and sex and adjusting for other clinical variables (severity of dementia ...) the patient's condition before and after admission, in terms of quality of life, dependency, instrumental activities of daily living and severity of dementia. 3. To compare the length of stay, complications, mortality rate, the degree of dependency and quality of life of patients with dementia compared to those without dementia, matched by groups of pathologies, gender and age.

ELIGIBILITY:
Inclusion Criteria:

* For the patients with dementia cohort, the inclusion criteria were: (a) Being patient aged over 75 years; (b) having been diagnosed with dementia according to the Diagnostic and Statistical Manual for Mental Disorders-IV (American Psychiatric Association, 1994) by any of the psychiatrists; (c) having received inpatient treatment by the time of the study in the hospital//with an unplanned medical admission to any medical speciality in the Galdakao-Usansolo Hospital (d) agreeing to participate voluntarily and providing written informed consent. Patients with dementia were included if a caregiver agreed to participate voluntarily. Caregiver is defined as any person who cares for a needy person in his or her direct environment on a regular basis and more or less as a matter of course. The caregiver is related (family, friend…) to the person receiving care and is not a professional caregiver (Shoenmakers et al., 2010).
* For the cognitive intact patients cohort, the inclusion criteria were patients without dementia admitted in the hospital by the time of the study, matched with patients with dementia, after controlling for age, gender and types of pathologies.

Exclusion Criteria:

* Patients with dementia (or caregivers) were excluded if they did not provide inform consent.
* The exclusion criteria for patients without dementia were disorders interfering with psychometric assessment, or not given written informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: For this prospective matched cohort study, the investigators recruited two groups of adults aged 75 years and older with an unplanned medical admission to any medical speciality between January 2012 and December 2014 in the Galdakao-Usansolo Hospital in the Basque Country (northern Spain), a 400-bed general teaching hospital serving a population of 300,000. It is one of the networks of public hospitals of the Basque Health Service, which provides free unrestricted care to nearly 100% of the population. One group (patients with dementia cohort) was drawn from patients with dementia, and a second group (patients without dementia cohort) of patients without dementia.
Sampling Method: Probability Sample
Enrollment: 413 (Actual)
Dates: Start 2012-01; Primary Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Mortality during hospitalization and at follow-up | Up to 3 months
  In-hospital mortality, and at follow-up: information on survival status of the patients was collected during hospitalization and assessed 3 months after discharge by telephone interview to patients or caregivers.

SECONDARY OUTCOMES:
The Alzheimer's Disease Test (AD8) | Up to 3 months
  The Alzheimer's Disease Test (AD8) is a brief informant-based measure that reliably distinguishes individuals with very mild dementia from those with normal cognition [Galvin et al., 2005). The AD8 is composed of 8 items. In the initial development of the AD8, using a cutoff of 2 or greater on the AD8 to predict dementia gave the most desirable combination of sensitivity (85%) and specificity (86%).
Assessment of Performance in Basic Activities of Daily Living: Barthel Index | Up to 3 months
  The Barthel Index is a scale used for the assessment of performance in basic activities of daily living [Mahoney & Barthel, 1965) that considers 10 basic functions and yields a score of 0-100. A higher score is associated with a greater likelihood of being able to live at home with a degree of independence following discharge from hospital. It was categorized according to four cutoff points, which are as follows: 75-100 as reference (no-mild disability), 50-74 (moderate disability), 25-49 (severe disability), and 0-24 (completely dependent).
Instrumental Activities of Daily Living (IADL) | Up to 3 months
  Lawton and Brody score was determined as a function of patient status 2 weeks before admission, based on the patient's medical history or information supplied by a caregiver. IADL assesses ability to use the telephone, to shop, to use transport, to cook, to do housework, to take medication and to handle finances. 0 indicates total dependence and the maximum score (8) indicates total independence.
EuroQoL 5-domain for Health-related quality of life (EQ-5D) (EuroQoL Group, 1990). | Up to 3 months
  This well-established generic instrument which measures health-related QoL has five domains: mobility, self-care, pain/discomfort, usual activities, and anxiety/depression. The respondents also rate their own health today on a visual analogue scale from 100 (best imaginable health state) to 0 (worst imaginable health state). The data can be presented descriptively as a health profile, and a single index utility score can be calculated.
The Quality of Life in Alzheimer's disease (QOL-AD) | Up to 3 months
  - The QOL-AD, a 13-item scale (range, 13 to 52, with higher scores indicating a better QOL) was used to examine AD-specific QOL (Logsdon et al., 1999). It has 13 items covering the domains of physical health, energy, mood, living situation, memory, family, marriage, friends, chores, fun, money, self, and life as a whole. These are scored on a 4-point Likert scale, ranging from 1 (poor) to 4 (excellent), with a possible total range from 13 to 52. The scale obtains separate ratings of the patient's QoL from both the patient and the caregiver, where available. These scores can be combined into a single score, weighting the person with dementia's own QoL score twice as heavily as the caregiver's. Early studies by Logsdon et al. (1999) suggest it to have good internal consistency, construct validity, and test-retest reliability. In this study, only the caregiver of the person with dementia's self-reported QoL was evaluated.
Caregiver's burden was evaluated with the Zarit Scale | Up to 3 months
  A reduced Zarit scale is useful to identify caregiver burden in dementias (with a sensitivity 98,5% and specificity of 94,7%), and it is also easy to use (Gort et al., 2010). Fields explored with the 4 items Zarit scale were overburden (items 9 and 14), irritability (item 5) and the self-care (item 2). These are scored on a 5-point Likert scale, ranging from 1 (never) to 4 (most times). Higher score, more burden. (in online material)
Diagnosis | Up to 3 months
Body Mass Index (BMI) | Up to 3 months
Nutritional status | Up to 3 months
  Blood test which included serum albumin, total cholesterol, electrolytes, total lymphocyte count was made.
Level of consciousness: The Glasgow Coma Scale (GCS) | Up to 3 months
  The Glasgow Coma Scale (GCS) was employed to measure consciousness (Teasdale & Jennett, 1974). In this scale the normal state merits a score of 15, and as level of consciousness deteriorates, the score becomes less. (Teasdale & Jennett, 1974).
Pressure Ulcer risk: the Braden Scale and the Gosnell Scale were employed. | Up to 3 months
  The Braden Scale (Bergstrom et al., 1987) is a summated rated scale comprised of 6 subscales: sensory perception, mobility, activity, moisture, nutrition, and friction and shear. The 6 subscales are rated from 1 to 4, except the friction and shear subscale, which is rated from 1 to 3. Each numerical rating has a definition of patient characteristics to evaluate when assigning a score. A total of 6 to 23 points is possible.

CONTACTS AND LOCATIONS:
Overall Officials: Inmaculada Moro, MSc, Principal Investigator — Hospital Galdakao-Usansolo